CLINICAL TRIAL: NCT03095326
Title: Pneumococcal Vaccination for Splenectomised Thalassemia Major Patients in Indonesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01
Record Dates: First submitted 2017-03-15; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Thalassemia; Pneumococcal Infection
MeSH Terms: conditions — Thalassemia; Pneumococcal Infections | interventions — Zinc; Zinc Sulfate; Sucrose; five-valent pneumococcal conjugate vaccine; 13-valent pneumococcal vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Intervention Model Description: All splenectomized thalassemia major subjects were provided with PCV pneumococcal vaccine (Prevenar 13®) at the start of the trial. The subjects were then randomly assigned into one of 2 groups (the zinc group and the placebo group). Zinc was provided in the form of syrup at a dose of 1.5 mg/kg/day, with a maximum of 50 mg/day. The placebo was also provided in the form of syrup, with similar shape and flavor.
Who Masked: Investigator
Masking Description: The participant are divided into two different groups, which are assigned with either zinc or placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc Syrup 1.5 mg/kgbw/day (Experimental): Patient were given zinc formula in the form of syrup with dosage of 1.5 mg/kg body weight/day with a maximum dose of 50 mg/day. The amount of syrup given is estimated to be enough for 4 weeks.
  Interventions: Dietary Supplement: Zinc; Biological: PCV Vaccine; Biological: PPV Vaccine
- Sucrose syrup (Placebo Comparator): Patient were given sucrose syrup as placebo. The syrup was made in the same flavor and consistency as the zinc syrup.
  Interventions: Drug: Sucrose; Biological: PCV Vaccine; Biological: PPV Vaccine

INTERVENTIONS:
Dietary Supplement: Zinc — formula of ZnSO4, usually used to treat zinc deficiency.
  Other Names: Zinc sulfate
  Arms: Zinc Syrup 1.5 mg/kgbw/day
Drug: Sucrose — Placebo of sucrose syrup
  Other Names: Sucrose syrup
  Arms: Sucrose syrup
Biological: PCV Vaccine — Pneumococcal conjugate vaccine
  Other Names: Prevenar 13®
Biological: PPV Vaccine — Pneumococcal polysaccharide vaccine
  Other Names: Pneumovax®

SUMMARY:
Splenectomized thalassemia major subjects were provided with PCV pneumococcal vaccine (Prevenar 13®) at the start of the trial, following which they were randomly assigned to 2 groups (zinc and placebo group). After 8 weeks, the subjects received PPV pneumococcal vaccine (Pneumovax®). Zinc syrup was provided to the zinc group at a dose of 1.5 mg/kg/day (maximum of 50 mg/day). Pneumococcal IgG examinations were conducted at the start of the trial and after 12 weeks.

DETAILED DESCRIPTION:
This study is a single blinded randomised-control trial. Splenectomized thalassemia major patient samples were provided with PCV pneumococcal vaccine (Prevenar 13®) at the start of the trial, following which they were randomly assigned to 2 groups (zinc and placebo group). After 8 weeks, the subjects received PPV pneumococcal vaccine (Pneumovax®). Zinc syrup was provided to the zinc group at a dose of 1.5 mg/kg/day (maximum of 50 mg/day). Placebo containing sucrose syrup of the same form, taste, consistency and color was given to the other group. Everyone except the primary researcher are blinded to which of the treatment is placebo and which is actual zinc syrup. Pneumococcal IgG examinations were conducted at the start of the trial and after 12 weeks.

Sample size was measured using:

n1=n2=n= {((Zα+Zβ) Sd)/d}^2 where N = number of subject Za = degree of significance (5%), a = 5% Zb = strength of study (80%). b = 20% Sd = standard deviation d = meaningful difference between the two groups The measured sample size is 816, but due to limited patient total population sampling was used instead.

ELIGIBILITY:
Inclusion Criteria:

* Splenectomised thalassemia patient

Exclusion Criteria:

* non-splenectomised thalassemia patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2014-02-01 (Actual)

PRIMARY OUTCOMES:
Pneumococcal IgG | week 12
  Pneumococcal IgG level was measured using Pneumococcus IgG Immunopotency

CONTACTS AND LOCATIONS:
Overall Officials: Teny T Sari, M.D, PhD, Principal Investigator — Faculty of Medicine University of Indonesia
Locations (1):
- Fakultas Kedokteran Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No